CLINICAL TRIAL: NCT05927506
Title: Adolescent Changes in Brain and Behavior in Boys and Girls With ADHD
Status: Completed | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00064633; IRB00064633 (Other: Johns Hopkins Hospital)
Record Dates: First submitted 2023-03-21; First posted 2023-07-03 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: Cognitive Testing; Typically Developing; Motor Control; Gender Differences
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents with ADHD: Observational study of behavior cognitive and motor control
  Interventions: Behavioral: Other
- Adolescents without ADHD: Observational study of behavior cognitive and motor control
  Interventions: Behavioral: Other

INTERVENTIONS:
Behavioral: Other — Observational study of behavior cognitive and motor control

SUMMARY:
The purpose of the study is to examine the developmental trajectory of response control in boys and girls with ADHD entering adolescence. The investigators also want to determine the developmental trajectory of brain anatomy and brain connectivity in boys and girls with ADHD entering adolescence.

DETAILED DESCRIPTION:
Children with Attention Deficit Hyperactivity Disorder (ADHD) are at risk for a host of deleterious outcomes including impaired social relations, academic difficulties, criminality, and comorbid psychopathology (substance use, depression, anxiety). Many of these difficulties emerge and exacerbate during adolescence; therefore, it is crucial to understand the developmental trajectory of ADHD-associated changes in brain and behavior during this sensitive period. Further, there is increasing recognition that sex may be an important moderator of the clinical manifestations of ADHD, with adolescent boys showing more impulsive risk-taking while girls show more emotional dysregulation.

Identification of patterns of brain and behavioral development associated with risk for poor outcome in both boys and girls with ADHD shows the profound public health significance of our research. Furthermore, the investigators are proposing to examine the dimensional construct of response control in children with ADHD from multiple levels of analysis including neural structure and connectivity, behavioral expression, and relation to functional outcomes, with the ultimate goal of identifying bio-behavioral markers of impairment and adjustment in children with ADHD.

Our objectives:

Aim 1: To examine the developmental trajectory of response control in boys and girls with ADHD entering adolescence.

Aim 2: To examine how baseline abnormalities in response control and brain structure and function, as well as development trajectories for these measures, differentially predict functional outcomes in adolescent boys and girls with ADHD.

Aim 3: To examine how intrinsic functional connectivity relates to brain structure, structural connectivity, and response control in adolescent boys and girls with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with or without Attention Deficit Hyperactivity Disorder
* Must be able to attend a follow-up after 18 months after initial visit

Exclusion Criteria:

* Diagnosed with Autism Spectrum Disorder (ASD)
* Diagnosed with Schizophrenia, Conduct Disorder, and/or Bipolar Disorder
* Diagnosed with a genetic disorder
* Premature birth (less than 36 weeks)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Male and Female adolescents within the age range of 12-17 years old, with or without a diagnosis of Attention Deficit Hyperactivity Disorder
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Response Control and Frustration Tolerance | Completed on Day 1 or Day 2 Visit
  Go/No-Go (GNG) reaction time task related to working memory and motivation. Each task will take place in a single block of 207 trials (80% green), with no rest phases (total duration = 8min, 19 sec). For the motivational GNG task, stimulus presentation will be followed by a blank screen (1000ms), the presentation of visual feedback (1700ms), and another blank screen (500ms). Reward feedback will be presented for correct "go" responses and response cost feedback will be presented for commission errors.
Developmental Trajectory of Brain Anatomy | Completed on Day 1 or Day 2 Visit
  The Primary outcome variables will be morphometry of cortical regions (thickness, surface area, folding index, volume) and subcortical regions (basal ganglia, amygdala, and hippocampus volume and shape).
Predictors of Adolescent Socio-Emotional Development | Completed on Day 1 or Day 2 Visit
  Behavior Assessment System for Children (BASC-3) is a questionnaire used to assess behavioral and emotional functioning in children. The parent-report, teacher-report, and self-report versions will be administered to collect behavioral and emotional values.
Developments of ADHD Symptoms | Completed on Day 1 or Day 2 Visit
  Conners-4 is a questionnaire to values on conduct and learning problems, impulsivity-hyperactivity, anxiety, and social competence. Parent-report and teacher-report will be administered collect values to determine ADHD symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Mostofsky, Ph.D, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Insititute, Baltimore, Maryland, United States